CLINICAL TRIAL: NCT00557349
Title: A Randomized, Double-blind Clinical Trial Comparing Zegerid Capsule to Famotidine in Preventing Anastomotic (Marginal) Ulcers in Post Gastric Bypass Patients
Brief Title: Ulcer Prevention Study in Post Gastric Bypass Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1058337
Record Dates: First submitted 2007-11-12; First posted 2007-11-14 (Estimated); Results first posted 2017-01-19 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2016-09

CONDITIONS: Marginal Ulcers
Keywords: gastric bypass surgery; anastomosis, Roux-en-Y; Complication, Postoperative
MeSH Terms: conditions — Peptic Ulcer; Postoperative Complications | interventions — Omeprazole; omeprazole, sodium bicarbonate drug combination; Famotidine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omeprazole (Active Comparator): 40 mg Omeprazole daily
  Interventions: Drug: Omeprazole
- Famotidine (Active Comparator): 40 mg Famotidine daily
  Interventions: Drug: Famotidine

INTERVENTIONS:
Drug: Omeprazole — 40mg dose administered as a suspension or capsule as physician directs daily at bedtime for 14 weeks beginning day of hospital discharge following gastric bypass surgery.
  Other Names: Zegerid
  Arms: Omeprazole
Drug: Famotidine — 40mg dose administered as a suspension or capsule as physician directs daily at bedtime for 14 weeks beginning day of hospital discharge following gastric bypass surgery.
  Other Names: Pepcid
  Arms: Famotidine

SUMMARY:
This research is to determine which medication, Zegerid (Omeprazole/Sodium Bicarbonate) or Pepcid AC (Famotidine), works best at reducing the chance that a patient will get an ulcer after gastric bypass surgery.

DETAILED DESCRIPTION:
The purpose of this research is to evaluate information about the control of gastric acid in post gastric bypass surgery patients. Goal is to determine which medication best reduces the incidence of anastomotic ulcers post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Subject is age ≥ 18 years
* Patient meets the criteria for laparoscopic gastric bypass surgery
* Females only: Patient is willing to take a urine pregnancy test

Exclusion Criteria:

* Subject allergic to omeprazole or famotidine
* Patient receiving antifungal (i.e. ketoconazole or itraconazole)
* Hepatic insufficiency
* History of Crohns disease
* History of Zollinger-Ellison disease
* Patient received an investigational drug within 30 days of enrollment
* Patient currently enrolled in another research project
* Females Only: Pregnancy or plan on becoming pregnant during the next 14 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-11; Primary Completion 2007-11 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger de la Torre, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri Health Care, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited from patients preparing for Roux-en-Y gastric bypass (RYGB) at Missouri Bariatric Services, the bariatric clinic associated with University of Missouri. Patients were recruited from November 2006 through November 2007.
Pre-assignment Details: While study participants were enrolled prior to their RYGB, they did not begin the study drug until after discharge from the hospital post-RYGB. During that time some patients were excluded, whether it was because the patient's surgery was cancelled or because the patient no longer met the inclusion/exclusion criteria.
Groups:
- Omeprazole; Famotidine: 40 mg daily at bedtime for 14 weeks
Period: Overall Study
Arm/Group | Omeprazole | Famotidine
Started | 22 (omeprazole/bicarb) | 18
Completed | 17 | 13
Not Completed | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Omeprazole; Famotidine: 40 mg daily for 14 weeks
- Total: Total of all reporting groups
Arm/Group | Omeprazole | Famotidine | Total
Number analyzed (Participants) | 22 | 18 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 18 | 40
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: participants] — Gender information is missing for the Famotidine arm.
  participants
    Unknown | 0 | 18 | 18
    Male | 8 | 0 | 8
    Female | 14 | 0 | 14
Region of Enrollment [Number; unit: participants]
  United States | 22 | 18 | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complaints, Specifically About Pain, Vomiting, Dyspepsia, and/or Dysphagia.
Time Frame: during first 14 weeks after surgery
Population: Patients lost to follow-up were not included in the data analysis.
Measure: Number; unit: participants
Arm/Group | Omeprazole | Famotidine
Number analyzed (Participants) | 17 | 13
participants | 17 | 13

2. Secondary Outcome: Number of Participants With Upper Endoscopy Indicated Due to Complaints
Description: Endoscopic visualization of presence or absence of anastomotic ulcers if upper endoscopy indicated due to patient complaints - based upon severity of complaints
Time Frame: during first 14 weeks after surgery
Population: Patients lost to follow-up were not included in the study analysis.
Measure: Number; unit: participants
Arm/Group | Omeprazole | Famotidine
Number analyzed (Participants) | 17 | 13
participants | 1 | 13

ADVERSE EVENTS:
Arm/Group | Omeprazole | Famotidine
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/13
Other Adverse Events (participants affected / at risk) | 0/17 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes